CLINICAL TRIAL: NCT00101998
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase IIb Study to Evaluate the Efficacy and Safety of Multiple Alvimopan Dosage Regimens for the Treatment of Opioid-Induced Bowel Dysfunction in Cancer Pain Subjects
Brief Title: Study Of Alvimopan Drug For Treatment Of Constipation Due To Prescription Pain Medication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3753-009; 767905/008 (Other: Cubist Study Number); NCT00903513 (obsolete NCT alias)
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Constipation; Bowel Dysfunction
Keywords: OBD (Induced Bowel Dysfunction); cancer pain; pain medication; constipation; bowel; bowel dysfunction
MeSH Terms: conditions — Constipation; Intestinal Diseases; Cancer Pain | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Alvimopan 0.5 mg Twice Daily (BID) (Experimental): 0.5 milligrams (mg) of alvimopan was administered orally BID for 3 weeks.
  Interventions: Drug: alvimopan
- Alvimopan 1 mg Once Daily (QD) (Experimental): 0.5 mg of alvimopan was administered orally QD for 3 days, then 1 mg of alvimopan QD for the remaining 3 weeks. Placebo was administered orally QD to maintain the blind.
  A protocol amendment dropped this arm because another study had demonstrated 1 mg QD treatment to have similar efficacy but a less favorable gastrointestinal-related safety profile compared with 0.5 mg BID treatment.
  Interventions: Drug: alvimopan; Drug: placebo
- Alvimopan 1 mg Twice Daily (BID) (Experimental): 0.5 mg of alvimopan was administered orally BID for 3 days, then 1 mg of alvimopan BID for the remaining 3 weeks.
  Interventions: Drug: alvimopan
- Placebo (Placebo Comparator): Placebo was administered orally BID for 3 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alvimopan
  Arms: Alvimopan 0.5 mg Twice Daily (BID); Alvimopan 1 mg Once Daily (QD); Alvimopan 1 mg Twice Daily (BID)
Drug: placebo
  Arms: Alvimopan 1 mg Once Daily (QD); Placebo

SUMMARY:
A multicenter study to evaluate the effectiveness and safety of multiple dosage regimens of an investigational drug for the treatment of constipation due to prescription pain medication in subjects with cancer pain. The study will require five visits over a five-week period.

ELIGIBILITY:
Inclusion criteria:

* Participant is in any stage of cancer but has a minimum life expectancy of at least 3 months at the time of the Screening Visit.
* Participant is taking opioid therapy for persistent cancer pain.
* Participant meets the definition of opioid-induced bowel dysfunction as follows: Since starting opioid therapy, the subject has had decreased bowel movement (BM) frequency and at least one of the following constipation symptoms [sensation of incomplete evacuation, difficulty in expelling stool (straining), hard stools (abnormal stool consistency)].
* Participant understands the procedures, agrees to participate in the study, and has signed and dated the informed consent form prior to the initiation of any study-related activities, including discontinuation of pre-study laxative regimen or other prohibited medications.
* Participant is able and willing to comply with a daily paper diary and is capable of completing paper questionnaires at study visits.

Exclusion criteria:

* Participant is pregnant or lactating, or planning to become pregnant.
* Participant is not ambulatory.
* Participant has participated in another trial with an investigational drug (unapproved), device or procedure within 30 days of the Screening Visit.
* Participant is unable to eat, drink, take/hold down oral medications.
* Participant is taking opioids for the management of drug addiction.
* Participant is unable or unwilling to discontinue the use of and/or refrain from using laxatives of all types and formulation at the Screening Visit and throughout the entire study.
* Participant has severe constipation that has not been appropriately managed such that the subject is at immediate risk of developing serious complications of constipation. This would include a subject who has reported no bowel movement for 7 consecutive days prior to the Screening Visit.
* Participant with gastrointestinal or pelvic disorders known to affect bowel transit, produce gastrointestinal (GI) obstruction, or contribute to bowel dysfunction.
* Participant is currently taking vinca alkyloids or plans to take vinca alkyloids during the study.
* Participant is currently undergoing abdominal radiation therapy and/or plans to undergo abdominal radiation therapy during the study.
* Participant is human immunodeficiency virus (HIV)-infected, has active hepatitis (any subtype including ongoing chronic hepatitis B), or has ever been infected with hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2006-05-01 (Actual); Study Completion 2006-05-01 (Actual)

PRIMARY OUTCOMES:
Change in weekly SCBM frequency. A SCBM is a spontaneous and complete bowel movement, which means a bowel movement that occurs with no laxative use in the prior 24 hours and leaves the subject with the feeling of complete evacuation of the rectum.

SECONDARY OUTCOMES:
Additional measures of Bowel movement (BM) frequency and symptoms, safety profile of the treatment regimens and any changes in pain intensity or opioid use.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (145):
- United States (61):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, La Verne, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Lecanto, Florida
  - GSK Investigational Site, Miami Shores, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Titusville, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Hutchinson, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Bethpage, New York
  - GSK Investigational Site, Huntington Station, New York
  - GSK Investigational Site, Jamaica, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Hendersonville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Middletown, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Portsmouth, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (2):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
- Australia (5):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Redcliffe, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Daw Park, South Australia
  - GSK Investigational Site, Malvern, Victoria
- Canada (13):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Chandler, Quebec
  - GSK Investigational Site, Lévis, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Québec
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- GSK Investigational Site, Helsinki, Finland
- France (3):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Villejuif
- Germany (2):
  - GSK Investigational Site, Goslar, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
- Hong Kong (3):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Zalaegerszeg-Pozva
- GSK Investigational Site, Bangalore, India
- Italy (11):
  - GSK Investigational Site, Caserta, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Forlì, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Busca (CN), Piedmont
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Florence, Tuscany
- GSK Investigational Site, Leeuwarden, Netherlands
- New Zealand (3):
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Hastings
  - GSK Investigational Site, Wellington
- GSK Investigational Site, Lahore, Pakistan
- GSK Investigational Site, Lima, Peru
- GSK Investigational Site, Manila, Philippines
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Otwock
  - GSK Investigational Site, Poznan
- GSK Investigational Site, Lisbon, Portugal
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, St'Petersburg
- South Africa (4):
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Groenkloof, Pretoria
  - GSK Investigational Site, Houghton, Johannesburg
  - GSK Investigational Site, Kenilworth, Cape Town
- GSK Investigational Site, Seoul, South Korea
- Spain (11):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sabadell / Barcelona
  - GSK Investigational Site, Serra / Valencia
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Soria
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Chiang Mai, Thailand
- United Kingdom (5):
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Surrey